CLINICAL TRIAL: NCT06407167
Title: Observational Cohort Study of the Neuropathic Pain in Surgical Treatment of Patients With Degenerative Lumbar Stenosis
Brief Title: Neuropathic Pain in Patients With Degenerative Lumbar Stenosis
Status: Active, not recruiting | Type: Observational
Sponsor: N.N. Priorov National Medical Research Center of Traumatology and Orthopedics (Other)
Responsible Party: Principal Investigator, Aleksandr Krutko, Head of Neurosurgery Department, N.N. Priorov National Medical Research Center of Traumatology and Orthopedics
Other Study IDs: NS12-02
Record Dates: First submitted 2024-04-24; First posted 2024-05-09 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Spinal Stenosis; Neuropathic Pain; Spinal Disease
MeSH Terms: conditions — Spinal Stenosis; Neuralgia; Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Neuropathic Pain: All patients will undergo lumbar decompression at stenosis levels (clinically and MRI confirmed) regardless of study group
  Interventions: Diagnostic Test: DN4 (Douleur Neuropathique 4 Questions) questionnaire
- No Neuropathic Pain: All patients will undergo lumbar decompression at stenosis levels (clinically and MRI confirmed) regardless of study group
  Interventions: Diagnostic Test: DN4 (Douleur Neuropathique 4 Questions) questionnaire

INTERVENTIONS:
Diagnostic Test: DN4 (Douleur Neuropathique 4 Questions) questionnaire — DN4 includes a series of ten questions consisting of both sensory descriptors and signs related to bedside sensory examination
  Other Names: neuropathic pain diagnostic questionnaire

SUMMARY:
Pre- and postoperative pain in patients with degenerative stenosis requires great attention, as it can mislead the doctor about treatment tactics. Neuropathic pain in the legs before and after the surgical procedure, as well as the residual or recurrent pain syndrome existing against this background, overshadow the patient's recovery and cast doubt on the fullness of the performed decompression. Neural compression in the spinal canal and back pain may be the cause of the patient's antalgic posture and sagittal imbalance as seen on X-Ray, to need for corrective interventions surgical procedure.

Thus, it is necessary to clarify the role and the influence of the pain and its type on the perioperative period in patients with degenerative lumbar spinal stenosis.

DETAILED DESCRIPTION:
The current study is prospective observational study to evaluate the role of pain syndrome including neuropathic pain in surgical outcomes in patients with degenerative lumbar spinal stenosis.

This study will be conducted at Priorov Central Institute for Trauma and Orthopedics, Moscow, Russia.

The study is expected to enroll at least 120 adult patients with degenerative lumbar stenosis. The neuropathy will be assessed preoperatively, and then the patient will undergo decompressive lumbar surgery without fusion.

The neuropathic pain will be evaluated according to DN4 preoperatively, each patient will be assigned to one of two groups depending on the total value of DN4 - with the presence of neuropathy (DN4>= 4) and without neuropathy (DN4 <4).

Postoperative evaluation will include 2 visits during one year to evaluate clinical and radiological outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years;
2. Radicular leg pain with or without neurogenic claudication with or without back pain;
3. Planned decompressive surgery for degenerative lumbar stenosis with or without degenerative spondylolisthesis;
4. Symptoms persisting for at least 3 months prior to surgery;
5. Given written Informed Consent;
6. Able and agree to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements

Exclusion Criteria:

1. Prior lumbar fusion at any level;
2. Any contraindication or inability to undergo baseline and/or follow up MRI or X-ray as required per protocol;
3. Back or non-radicular pain of unknown etiology;
4. History or presence of any other major neurological disease or condition that may interfere with the study assessments (e.g. significant peripheral neuropathy, multiply sclerosis);
5. Any other condition or situation that the investigator believes may interfere with the safety of the subject or the intent and conduct of the study;
6. Previous enrollment in this study, current enrollment or plans to be enrolled in another study (in parallel to this study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One study center in Russia will include adult patients with radicular leg pain with/without neurogenic claudication with/without back pain caused by degenerative spinal stenosis with MRI-confirmed nerve compression; with symptoms persisting for more than 3 months before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Oswestry Disability Index (ODI) | 3 months postoperatively
  To observe the change of Oswestry Disability Index as compared to baseline through follow-up terms

SECONDARY OUTCOMES:
Change from baseline in Neuropathic Pain 4 Questions (DN4) | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the change of Neuropathic Pain 4 Questions as compared to baseline through follow-up terms
Change from baseline in Numeric Pain Rating Scale (NPRS) | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the change of Numeric Pain Rating Scale as compared to baseline through follow-up terms
Change from baseline in Oswestry Disability Index (ODI) | 12 months postoperatively
  To observe the change of Oswestry Disability Index as compared to baseline through follow-up terms
Change from baseline in The Health Transition Item from SF-36 (HTI Item) | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the change of The Health Transition Item as compared to baseline through follow-up terms
Change from baseline in sagittal balance parameters | 3 months, 12 months postoperatively
  To observe the change of sagittal balance parameters (index Barrey) as compared to baseline through follow-up terms
Change from baseline in regional balance parameters | 3 months, 12 months postoperatively
  To observe the change of regional balance parameters (Segmental Lordosis) as compared to baseline through follow-up terms
Change from baseline in frontal balance parameters | 3 months, 12 months postoperatively
  To observe the change of frontal balance parameters (Cobb's angle) as compared to baseline through follow-up terms
the safety parameters | during study, an average of 1 year
  To observe and document the safety parameters (Adverse events)

CONTACTS AND LOCATIONS:
Locations (1):
- Priorov National Medical Research Center of Traumatology and Orthopedics, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No